CLINICAL TRIAL: NCT03018730
Title: An Open Label Study of the Safety and Efficacy of PRX-102 in Patients With Fabry Disease Currently Treated With REPLAGAL® (Agalsidase Alfa)
Brief Title: Safety and Efficacy of PRX-102 in Patients With Fabry Disease Currently Treated With REPLAGAL® (Agalsidase Alfa)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Protalix (Industry)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB-102-F30
Record Dates: First submitted 2017-01-09; First posted 2017-01-12 (Estimated); Results first posted 2022-06-29 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Fabry Disease
Keywords: Fabry disease; Enzyme-Replacement Therapy; pegunigalsidase alfa; PRX-102; alpha galactosidase-A
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRX-102 (Experimental): PRX-102 infusion every 2 weeks
  Interventions: Biological: PRX-102 (pegunigalsidase alfa)

INTERVENTIONS:
Biological: PRX-102 (pegunigalsidase alfa) — PRX-102 1 mg/kg every 2 weeks
  Other Names: pegunigalsidase alfa; Recombinant human alpha galactosidase-A

SUMMARY:
This is an open label switch over study to assess the safety and efficacy of PRX-102 (pegunigalsidase alfa). Patients treated with agalsidase alfa for at least 2 years and on a stable dose (>80% labelled dose/kg) for at least 6 months. Patients will be screened and evaluated over 3 months while continuing on agalsidase alfa. Following the screening period, the patient will be enrolled and switched from their agalsidase alfa treatment to receive intravenous (IV) infusions of PRX-102 1 mg/kg every two weeks for 12 months. No more than 25% of treated patients will be female.

DETAILED DESCRIPTION:
Dosage and administration details:

pegunigalsidase alfa individual dose for each patient was prepared according to the patient's weight. Pegunigalsidase alfa administrated at 1 mg/kg, intravenously over 3 hours, every 2 weeks. After the first 2 months of treatment with pegunigalsidase alfa, infusion time may be reduced gradually to 1.5 hours pending patient tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-60 years
2. A documented diagnosis of Fabry disease
3. Males: plasma and/or leucocyte alpha galactosidase activity (by activity assay) less than lower limit of normal according to laboratory range and one or more of the characteristic features of Fabry disease i. Neuropathic pain ii. Cornea verticillata iii. Clustered angiokeratoma
4. Females: historical genetic test results consistent with Fabry mutations, or in the case of novel mutations a first degree male relative with Fabry disease, and one or more of the characteristic features of Fabry disease i. Neuropathic pain ii. Cornea verticillata iii. Clustered angiokeratoma
5. Treatment with agalsidase alfa for at least 2 years and on a stable dose (>80% labelled dose/kg) for at least 6 months
6. eGFR ≥ 40 ml/min/1.73 m2 by CKD-EPI equation
7. Availability of at least 2 historical serum creatinine evaluations since starting agalsidase alfa treatment and not more than 2 years
8. Female patients and male patients whose co-partners are of child-bearing potential agree to use a medically acceptable method of contraception, not including the rhythm method

Exclusion Criteria:

1. History of anaphylaxis or Type 1 hypersensitivity reaction to agalsidase alfa
2. History of renal dialysis or transplantation
3. History of acute kidney injury in the 12 months prior to screening, including specific kidney diseases (e.g., acute interstitial nephritis, acute glomerular and vasculitic renal diseases); non-specific conditions (e.g, ischemia, toxic injury); as well as extrarenal pathology (e.g., prerenal azotemia, and acute postrenal obstructive nephropathy)
4. Angiotensin converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) therapy initiated or dose changed in the 4 weeks prior to screening
5. Urine protein to creatinine ratio (UPCR) > 0.5 g/g and not treated with an ACE inhibitor or ARB
6. Known history of hypersensitivity to Gadolinium contrast agent that was not managed by the use of premedication;
7. Females who are pregnant, planning to become pregnant during the study, or are breast feeding
8. Cardiovascular event (myocardial infarction, unstable angina) in the 6 month period before screening
9. Congestive heart failure NYHA Class IV
10. Cerebrovascular event (stroke, transient ischemic attack) in the 6 month period before screening
11. Presence of any medical, emotional, behavioral or psychological condition that, in the judgment of the Investigator and/or Medical Monitor would interfere with the patient's compliance with the requirements of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2020-01-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- Royal Melbourne Hospital, Parkville, Victoria, Australia
- Capital Health, Halifax, Nova Scotia, Canada
- Vseobecna fakultni nemocnice v Praze, Prague, Czechia
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Helse Bergen HF Haukeland Universitetssykehus, Bergen, Norway
- General Hospital Slovenj Gradec, Slovenj Gradec, Slovenia
- United Kingdom (3):
  - Queen Elizabeth Hospital, Department of Neurology,, Edgbaston, Birmingham
  - The Royal Free Hospital, London
  - Salford Royal NHS Foundation Trust, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azimpour K, Dorling P, Koulinska I, Kunduri S, Lan Z, Poritz J, Tremblay G, Raad-Faherty A. Health State Utility Values in Fabry Disease: Insights from the Pegunigalsidase Alfa Clinical Trials. Adv Ther. 2025 Mar;42(3):1421-1434. doi: 10.1007/s12325-024-03095-2. Epub 2025 Jan 23. PMID 39847314
- [Derived] Linhart A, Dostalova G, Nicholls K, West ML, Tondel C, Jovanovic A, Giraldo P, Vujkovac B, Geberhiwot T, Brill-Almon E, Alon S, Chertkoff R, Rocco R, Hughes D. Safety and efficacy of pegunigalsidase alfa in patients with Fabry disease who were previously treated with agalsidase alfa: results from BRIDGE, a phase 3 open-label study. Orphanet J Rare Dis. 2023 Oct 21;18(1):332. doi: 10.1186/s13023-023-02937-6. PMID 37865771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 22 adult patients were planned to be included in the study; no more than 25% were planned to be female patients. In practice, 15 males and 7 females (32%) received treatment in this study; 20 patients (13 males and 7 females) completed the 12 month treatment duration.
Groups:
- PRX-102: PRX-102 (pegunigalsidase alfa): PRX-102 infusion 1 mg/kg every 2 weeks
Period: Overall Study
Arm/Group | PRX-102
Started | 22
Completed | 20
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- PRX-102: PRX-102 infusion 1 mg/kg every 2 weeks
Arm/Group | PRX-102
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 0
  Race: Black or African American | 0
  Race: Native Hawaiian or other Pacific Islander | 0
  Race: White | 22
Region of Enrollment [Number; unit: participants]
  Canada | 2
  Netherlands | 1
  Czechia | 8
  Norway | 2
  United Kingdom | 6
  Slovenia | 1
  Australia | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.03
Description: Results represent the number of treatment-emergent adverse events (TEAE) that were considered possibly, probably, or definitely related to treatment
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | PRX-102
Number analyzed (Participants) | 22
participants
  At least 1 TEAE | 21
  At least 1 mild or moderate TEAE | 19
  At least 1 severe TEAE | 4
  At least 1 SAE | 4
  At least 1 TEAE unrelated or unlikely related | 19
  At least 1 TEAE related to study treatment | 5
  At least 1 SAE related to study treatment | 2
  At least 1 TEAE leading to discontinuation | 2
  At least 1 TEAE leading to death | 0

2. Other Pre Specified Outcome: eGFR
Description: eGFR was calculated based on the serum creatinine values that were assessed at weeks 4, 8, 12, 16, 20, 26, 30, 34, 38, 42, 46, 52 according to the CKD-EPI formula, baseline and Month 12 (week 52) reported. The absolute change in eGFR from baseline measurement at visit 1 prior to first PRX-102 infusion to last measurement at Month 12 was summarized using descriptive statistics.
Time Frame: Baseline and Month 12 (week 52)
Measure: Mean (Standard Error); unit: mL/min/1.73m^2
Groups:
- PRX-102 Efficacy Population; PRX-102 Male; PRX-102 Female: PRX-102 infusion 1 mg/kg every 2 weeks
Arm/Group | PRX-102 Efficacy Population | PRX-102 Male | PRX-102 Female
Number analyzed (Participants) | 20 | 13 | 7
mL/min/1.73m^2
  Baseline eGFR | 79.46 (4.92) | 75.87 (6.62) | 86.14 (6.72)
  Month 12 (week 52) eGFR | 76.91 (5.22) | 74.27 (7.15) | 81.80 (7.09)
  Change in eGFR from Baseline to Month 12 (week 52) | -2.56 (2.14) | -1.60 (2.75) | -4.34 (3.54)

3. Other Pre Specified Outcome: Mean Annualised Change in eGFR (Slope)
Description: The annualized change in eGFR (slope) per patient was calculated with all available eGFR values using a linear regression.
  The mean pre-switch slope is the eGFR slope during screening period and pre-infusion visit 1 (while on Replagal®).
  The mean post-switch slope is the eGFR slope during PRX-102 treatment, calculated based on eGFR vales at weeks 4, 8, 12, 16, 20, 26, 30, 34, 38, 42, 46, 52 after visit 1.
  The mean change in eGFR slope from pre- to post-switch is the mean difference between the two slopes.
  eGFR was calculated based on the serum creatinine values according to the CKD-EPI formula.
Time Frame: Pre-switch, Post-switch
Measure: Mean (Standard Error); unit: mL/min/1.73m^2/year
Arm/Group | PRX-102 Efficacy Population | PRX-102 Male | PRX-102 Female
Number analyzed (Participants) | 20 | 13 | 7
mL/min/1.73m^2/year
  pre-switch | -5.9 (1.34) | -6.36 (1.89) | -5.03 (1.65)
  post-switch | -1.19 (1.77) | -1.73 (2.64) | -0.21 (1.47)
  Change in eGFR slope from pre- to post-switch | 4.70 (2.26) | 4.63 (3.48) | 4.83 (1.09)

4. Other Pre Specified Outcome: Plasma Lyso-Gb3
Description: Plasma Lyso-Gb3 is Fabry disease specific biomarker that can assess treatment outcome which was measured at Baseline and weeks 12, 26, 38, 52. Baseline and Month 12 (week 52) reported.
Time Frame: Baseline and month 12 (week 52)
Measure: Mean (Standard Error); unit: nM
Arm/Group | PRX-102 Efficacy Population | PRX-102 Male | PRX-102 Female
Number analyzed (Participants) | 20 | 13 | 7
nM
  Baseline | 38.51 (9.68) | 51.81 (13.60) | 13.81 (2.31)
  Month 12 (Week 52) | 24.20 (5.10) | 32.25 (6.89) | 9.24 (1.08)
  Change from Baseline | -14.31 (5.13) | -19.55 (7.55) | -4.57 (1.42)

5. Other Pre Specified Outcome: Number of Participants According to Protein/Creatinine Ratio (UPCR)
Description: Urine Protein to Creatinine Ratio (UPCR), assessed by spot urine test, at Month 12 (Week 52).Number of Participants According to Protein/Creatinine Ratio (UPCR) level
Time Frame: 12 months
Measure: Number; unit: Subjects
Arm/Group | PRX-102 Efficacy Population | PRX-102 Male | PRX-102 Female
Number analyzed (Participants) | 20 | 13 | 7
Subjects
  Protein Undetectable | 9 | 7 | 2
  Normal to Mildly increased | 4 | 2 | 2
  Moderately increased | 2 | 0 | 2
  Severely increased | 5 | 4 | 1

6. Other Pre Specified Outcome: Left Ventricular Mass Index (g/m^2) by MRI
Description: Left ventricular mass was determined based on cardiac MRI data and the LVMI was indexed to patient's body surface area (g/m^2). In male patients the normal range for LVMI was 57-91 g/m^2, in female patients 47-77 g/m^2.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: g/m^2
Arm/Group | PRX-102 Efficacy Population | PRX-102 Male | PRX-102 Female
Number analyzed (Participants) | 20 | 13 | 7
g/m^2
  Baseline | 86.9 (6.9) | 97.6 (8.9) | 66.9 (5.8)
  Month 12 (Week 52) | 89.4 (6.1) | 98.3 (7.8) | 74.1 (7.2)
  Change from Baseline | 4.1 (2.8) | 2.4 (3.4) | 7.1 (5.0)

7. Other Pre Specified Outcome: Quality of Life EQ VAS
Description: The EQ VAS, of the EQ 5D 5L questionnaire, records the subject's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' (score "100") and 'Worst imaginable health state' (score "0").
Time Frame: 12 months
Measure: Mean (Standard Error); unit: Score
Arm/Group | PRX-102 Efficacy Population | PRX-102 Male | PRX-102 Female
Number analyzed (Participants) | 20 | 13 | 7
Score
  Baseline | 71.8 (4.3) | 66.8 (5.3) | 81.6 (6.1)
  Month 12 | 76.9 (4.5) | 71.5 (5.4) | 86.7 (7.0)
  Change from Baseline | 5.1 (3.3) | 4.8 (4.9) | 5.6 (3.0)

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- All Patients: PRX-102 infusion 1 mg/kg every 2 weeks
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 4/22
Other Adverse Events (participants affected / at risk) | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=22)
Type I hypersensitivity (Immune system disorders) | 2
Infectious mononucleosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=22)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3)
Palpitations (Cardiac disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Type 1 hypersensitivity (Immune system disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (5)
Dizziness (Nervous system disorders) | 2 (8)
Fatigue (General disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 2 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 7 (9)
Lower respiratory tract infection (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial agreement that is generally provided to the sites and Investigators contains a Publication paragraph that indicates the following: shall not, without the Sponsor's prior written consent, independently publish, present or otherwise disclose any results of or information pertaining to the trial until a multi-center publication is published, subject to certain limitations regarding timing and the confidentiality of unpublished data.

DOCUMENTS (2):
  • Study Protocol (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/30/NCT03018730/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT03018730/SAP_001.pdf